CLINICAL TRIAL: NCT04810416
Title: Effect of Texting and Writing on Hand Grip and Key Pinch Strength Among Collegiate Students
Brief Title: Effect of Texting and Writing on Grip and Pinch Strength
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Collaborators: King Saud University (Other)
Responsible Party: Principal Investigator, Tarek Mohamed El-gohary, Associate Professor, General Committee of Teaching Hospitals and Institutes, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CMR-PT-2021-09
Record Dates: First submitted 2021-03-12; First posted 2021-03-23 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Muscle Weakness Condition; Hand Grasp
Keywords: Hand grip strength, key pinch, risk factors, students; Key pinch; Risk factors; Students

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the parallel four groups
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessor will be masked to the participant's assigned activity and participants will be masked to the exact outcome measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Texting- 10 minutes (Experimental): Assigned participants will do texting for 10 minutes.
  Interventions: Other: Texting- 10 minutes
- Writing- 10 minutes (Experimental): Assigned participants will do writing for 10 minutes.
  Interventions: Other: Writing- 10 minutes
- Texting- 15 minutes (Experimental): Assigned participants will do texting for 15 minutes.
  Interventions: Other: Texting- 15 minutes
- Writing-15 minutes (Experimental): Assigned participants will do writing for 15 minutes.
  Interventions: Other: Writing- 15 minutes
- Control group (No Intervention): No hand activities.

INTERVENTIONS:
Other: Texting- 10 minutes — Participants will practice texting for 10 minutes using smart phone.
  Arms: Texting- 10 minutes
Other: Writing- 10 minutes — Participants will practice writing on notebook for 10 minutes.
  Arms: Writing- 10 minutes
Other: Texting- 15 minutes — Participants will practice texting for 15 minutes using smart phone.
  Arms: Texting- 15 minutes
Other: Writing- 15 minutes — Participants will practice writing on notebook for 15 minutes.
  Arms: Writing-15 minutes

SUMMARY:
Texting and writing are common hand activities among college students. Students tend to spend increasing hours of texting and writing for every day activities in addition to the academic assignments that are mainly on line and through distance education. The effect of such daily activities on hand grip and key pinch strength has not been studied among college students.

DETAILED DESCRIPTION:
Students will be recruited from physical therapy department of college of medical rehabilitation sciences after satisfying the inclusion and exclusion criteria. Participants will be randomly assigned to one of the four groups (texting 10 minutes, texting 15 minutes, writing 10 minutes and writing 15 minutes). Participants will be blinded to the outcome measures and the evaluator will be blinded to the participants assigned group. Hand grip strength and key pinch strength will be the main outcome measures. Participants demographics will be gathered in addition to recreational status, risk factors, pain body diagram and number of hours spent for texting and writing in every day life.

ELIGIBILITY:
Inclusion Criteria:

* Active college student
* Healthy
* Willing to participate
* Using smart phones& electronics
* Hand writing for > 10 minutes/day

Exclusion Criteria:

* Recent upper limbs injury (sprain& strain)
* Chronic neurological disorder
* Carpal tunnel syndrome
* De Quervain's disease
* Diabetic neuropathy

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Hand grasp Hand grasp | Up to 12 weeks
  Grip strength of the right- hand dominant will be measured at two wrist positions.
Key pinch | Up to 12 weeks
  Key pinch strength of the right- hand dominant will be measured.

SECONDARY OUTCOMES:
Borg CR-10 | Up to 12 weeks
  Rating the perceived exertion just after hand activity session.

CONTACTS AND LOCATIONS:
Locations (2):
- Saudi Arabia (2):
  - College of Medical Rehabilitation Sciences, Madinah
  - College of medical rehabilitation sciences, Madinah

IPD SHARING:
Plan to Share IPD: No
Hand grip and key pinch strength outcome measures will be shared.

REFERENCES:
- [Derived] Fathi El-Gohary TM, Aljohani MM. Effect Of Texting And Handwriting On Hand-Grip And Key-Pinch Strength Among Female-Collegiate Students: Randomized Controlled Trial. J Pak Med Assoc. 2023 Aug;73(8):1577-1582. doi: 10.47391/JPMA.1577. PMID 37697745